CLINICAL TRIAL: NCT06345534
Title: Randomized Comparison Between the FAST-FORWARD Schedule and the HAI5 Schedule for Breast Cancer Radiotherapy in 5 Fractions
Brief Title: FAST-FORWARD vs HAI5
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0255
Record Dates: First submitted 2024-03-14; First posted 2024-04-03 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Cancer, Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Intervention Model Description: Patients participating in the study will be randomized 1:1 between the FAST-FORWARD schedule and the HAI5 schedule. The first group is treated according to the FAST-FORWARD schedule, consisting of 5 radiation sessions on 5 consecutive working days (e.g. Monday to Friday). 2 rest days are allowed in the schedule, so that the treatment lasts a maximum of 7 days. The second group is treated according to the HAI5 schedule, developed by the radiotherapy department of Ghent University Hospital. In this schedule, at least 1 day of rest is scheduled between each treatment session, so the treatment is administered over 10-14 days.
Masking Description: Both healthcare provider and patient know the treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAST-FORWARD schedule (Other): The first group is treated according to the FAST-FORWARD schedule, consisting of 5 radiation sessions on 5 consecutive working days (e.g. Monday to Friday). 2 rest days are allowed in the schedule, so that the treatment lasts a maximum of 7 days.
  Interventions: Device: Questionnaire
- HAI5 schedule (Other): The second group is treated according to the HAI5 schedule, developed by the radiotherapy department of Ghent University Hospital. In this schedule, at least 1 day of rest is scheduled between each treatment session, so the treatment is administered over 10-14 days.
  Interventions: Device: Questionnaire

INTERVENTIONS:
Device: Questionnaire — Patients will be asked to complete questionnaires at different times (before, during and after radiation) to evaluate which schedule gives the fewest side effects and the best quality of life.
  The basic questionnaire and questionnaire about early side effects will be completed weekly up to 6 weeks after radiotherapy. The questionnaire about late side effects will be completed: after 6 months, 1 year, 2 years, 3 years, 4 years and 5 years.

SUMMARY:
Randomized comparison between the FAST-FORWARD schedule and the HAI5 schedule for breast cancer radiotherapy in 5 fractions.

DETAILED DESCRIPTION:
Previously, radiotherapy treatments for breast cancer usually consisted of 20-25 sessions to treat the entire breast, followed by an additional dose ("boost") to the tumor bed of 4-8 sessions. Today, 15-16 treatment sessions have become standard for whole breast irradiation, followed by a boost if indicated. The durability of further shortening the treatment to 5 sessions was proven in the FAST and FAST-FORWARD studies. After 10 and 5 years, the outcome was comparable with 25 and 15 radiation sessions, both in terms of toxicity and locoregional control.

There are currently 2 radiotherapy schedules in 5 sessions in use in Belgium (the FAST-FORWARD schedule and the HAI5 schedule), both of which have their advantages and disadvantages. In this project we want to investigate which schedule gives the fewest side effects and the best quality of life using questionnaires at different times (before, during and after radiation).

Patients participating in the study will be randomized 1:1 between the FAST-FORWARD schedule and the HAI5 schedule. The first group is treated according to the FAST-FORWARD schedule, consisting of 5 radiation sessions on 5 consecutive working days (e.g. Monday to Friday). In the schedule 2 rest days are allowed, so that the treatment lasts a maximum of 7 days. The second group is treated according to the HAI5 schedule, developed by the radiotherapy department of Ghent University Hospital. In this schedule, at least 1 day of rest is scheduled between each treatment session, so the treatment is administered over 10-14 days.

ELIGIBILITY:
Inclusion Criteria:

* histopathological diagnosis of breast cancer
* age 18 years or older
* male or female
* treated with breast conserving surgery or mastectomy with curative intent
* multidisciplinary decision of adjuvant radiotherapy after surgery

Exclusion Criteria:

* distant metastases
* decision of preoperative radiotherapy
* decision of partial breast irradiation
* positive resection margins ('ink on tumour')
* indication for boost on lymph node(s)
* history of thoracic or ipsilateral axillary radiotherapy (including radiotherapy of the contralateral breast or chest wall)
* need for bilateral irradiation
* breast reconstruction or expander
* patients unlikely to comply with the protocol (e.g. inability or unwillingness to complete the questionnaires at different time points).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Early side effects | Weekly up to 6 weeks after radiotherapy
  To evaluate radiotherapy-related symptoms in the chest/chest wall weekly up to 6 weeks after radiotherapy, evaluated with the standardized EORTC QLQ-BR23 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Liv Veldeman, MD, PhD, Principal Investigator — UZ Ghent
Locations (2):
- Belgium (2):
  - Universitary Hospital, Ghent
  - University Hospital Ghent, Ghent